CLINICAL TRIAL: NCT03803059
Title: A Single-Center Trial to Evaluate the Efficacy and Tolerability of SkinPen on Male and Female Subjects' Wrinkles of the Neck
Brief Title: Efficacy and Tolerability of SkinPen on Male and Female Subjects' Wrinkles of the Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bellus Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bellmed002
Record Dates: First submitted 2019-01-09; First posted 2019-01-14 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-07

CONDITIONS: Wrinkles

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Wrinkles of the Neck (Experimental): Microneedle treatment neck areas.
  Interventions: Device: SkinPen Precision

INTERVENTIONS:
Device: SkinPen Precision — Surgical instrument motors and accessories/attachments/Hydrogel

SUMMARY:
This single-center, the clinical trial is being conducted over the course of 90 days followed by 1-month and 6-month post-treatment visits in order to assess the efficacy and tolerability of the Sponsor's SkinPen device when used by men and women with the wrinkles of the neck.

DETAILED DESCRIPTION:
A total of 32 subjects completed study participation.

At visit 1 (baseline), subjects were screened for eligibility criteria, and those who qualified either completed day 1 procedures at the same visit or returned to the clinic up to 14 days after visit 1 to complete day 1 procedures at visit 2.

On days 1, 30, 60, and 90, after completion of visit assessments, doctors or fellows at the testing facility (henceforth referred to as "clinic") treated each subject's wrinkles of the neck with SkinPen Precision System at depths of up to 2.5mm.

During the post-treatment period, Clinical evaluations were conducted at visit 2 (day 1), visit 3 (day 30), visit 4 (day 60), visit 5 (day 90), visit 6 (1month post-treatment), and visit 7 (3 months post-treatment)

ELIGIBILITY:
Inclusion Criteria:

At least 20% of subjects will have Fitzpatrick skin types IV-VI Individuals who grade a 4 or higher on the Fitzpatrick Wrinkle Scale Individuals that desire correction of their wrinkles Individuals willing to withhold aesthetic therapies to the areas of the neck being treated or judged to potentially impact results by the Investigator.

Women of childbearing potential agree to take a urine pregnancy test at the Baseline visit and 6-months post-treatment or when deemed by Investigator and/or Sponsor. This may be changed to one monthly pregnancy test at the Sponsor's discretion. Women who are of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the baseline visit. Women must be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

* Postmenopausal for at least 12 months prior to the study;
* Without a uterus and/or both ovaries;
* Bilateral tubal ligation at least 6 months prior to study enrollment. Women of child bearing potential agree to take a urine pregnancy test at the Baseline visit and 6-months post-treatment or when deemed by Investigator and/or Sponsor. This may be changed to one month pregnancy test at the Sponsor's discretion. Women who are of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the baseline visit. Women must be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:
* Postmenopausal for at least 12 months prior to the study;
* Without a uterus and/or both ovaries;
* Bilateral tubal ligation at least 6 months prior to study enrollment.

Individuals of child-bearing potential who use an acceptable method of contraception throughout the study. Acceptable methods of birth control include:

1. Established use of hormonal methods of contraception (oral, injected, implanted, patch, or vaginal ring).
2. Barrier methods of contraception with spermicide: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
3. Intrauterine device (IUD) or intrauterine system (IUS)
4. Surgical sterilization (e.g., vasectomy that has been confirmed effective by sperm count check, tubal occlusion, hysterectomy, bilateral salpingectomy/oophorectomy)
5. Abstinence from heterosexual intercourse, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

   * Individuals that are willing to provide written informed consent and are able to read, speak, write, and understand English.
   * Individuals willing to sign a photography release.
   * Willingness to cooperate and participate by following study requirements (including those outlined in section 5.5) for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.

   Exclusion Criteria:
   * Individuals diagnosed with known allergies to facial or general skincare products.
   * Individuals who have the presence of an active systemic or local skin disease that may affect wound healing.
   * Individuals who have severe solar elastosis.
   * Individuals with sensitivity to topical lidocaine.
   * Individuals who have physical or psychological conditions unacceptable to the Investigator.
   * Individuals who have a recent history of significant trauma to the areas to be treated (< 6 months).
   * Individuals who have significant scarring, other than acne scars, in the area(s) to be treated.
   * Individuals who have severe or cystic active and clinically significant acne on the area(s) to be treated. Clinically significant acne is defined as a subject who has > 5 active inflammatory acne lesions (including acne conglobate, nodules, or cysts) in either the right or left treatment area.
   * Individuals who have a recent or current history of inflammatory skin disease, infection, cancerous/pre-cancerous lesion, unhealed wound or clinically significant acne in the proposed treatment areas. Individuals who have a history of systemic granulomatous diseases, active or inactive, (e.g. Sarcoid, Wegeners, TB, etc.) or connective tissue diseases (e.g. lupus, dermatomyositis, etc.).
   * Individuals who currently have or have a history of hypertrophic scars or keloid scars.
   * Individuals who currently have cancerous or pre-cancerous lesions in the areas to be treated and/or with a history of skin cancer.
   * Individuals who have the inability to understand instructions or to give informed consent.
   * Individuals who have had microdermabrasion or glycolic acid treatment to the treatment area(s) within 1 month prior to study participation or who will have this treatment during the study.
   * Individuals who have a history of chronic drug or alcohol abuse.
   * Individuals undergoing concurrent therapy that, in the Investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
   * Individuals who, in the Investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
   * Individuals who are current smokers or have smoked in the last 5 years.
   * Individuals who have a history of the following cosmetic treatments in the area(s) to be treated:

     * Skin tightening procedure within the past year;
     * Injectable filler of any type within the past:

       * 12 months for Hyaluronic acid fillers (e.g. Restylane)
       * 12 months for Ca Hydroxyapatite fillers (e.g. Radiesse)
       * 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra)
       * Ever for permanent fillers (e.g. Silicone, ArteFill)
     * Neurotoxins within the past 3 months;
     * Ablative resurfacing laser treatment;
     * Non-ablative, rejuvenating laser or light treatment within the past 6 months;
     * Surgical dermabrasion or deep facial peels;
     * Had a chemical peel, dermabrasion, non-ablative laser, or fractional laser resurfacing of the neck within 4 weeks
   * Individuals with a history of using the following prescription medications:

     * Accutane or other systemic retinoids within the past 6 months;
     * Topical Retinoids within the past 2 weeks;
     * Prescription-strength skin lightening devices (e.g. hydroquinone, tretinoin, AHA, BHA and polyhydroxy acids, 4-hydroxyanisole alone or in combination with tretinoin, etc.) within 4 months;
     * Any anti-wrinkle, skin lightening devices, or any other device or topical or systemic medication is known to affect skin aging or dyschromia (devices containing alpha/beta/poly-hydroxy acids, vitamin C, soy, Q-10, hydroquinone; systemic or licorice extract (topically), Tego® Cosmo C250, Giga white, lemon juice extract (topically), Emblica extract, etc.) within 2 weeks;
     * Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix, chronic NSAID use); and/or
     * Psychiatric drugs that in the Investigator's opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.
   * Individuals who are nursing, pregnant, or planning to become pregnant during the study according to the subject self-report.
   * Individuals having a health condition and/or pre-existing or dormant dermatologic disease on the face or body (e.g., psoriasis, rosacea, eczema, seborrheic dermatitis, vitiligo, hyper or hypo-skin pigmentation conditions such as post-inflammatory hyperpigmentation) that the Investigator or designee deems inappropriate for participation or could interfere with the outcome of the study.
   * Individuals with a history of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation as determined by study documentation.
   * Individuals with uncontrolled diseases such as asthma, diabetes, hyperthyroidism, medically significant hypertension or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
   * Individuals with any planned surgeries, overnight hospitalization, and/or invasive medical procedures during the course of the study.
   * Individuals who are currently participating in any other study involving the use of investigational devices or drugs or have participated in any clinical trial at UT Southwestern or at another research facility or doctor's office within 4 weeks prior to inclusion into the study.
   * Individuals who have an observable suntan, nevi, excessive hair, etc. or other dermal conditions on the neck that might influence the test results in the opinion of the Investigator or designee.
   * Individuals who have any condition, which in the opinion of the Investigator makes the patient unable to complete the study per protocol (e.g. patients not likely to avoid other facial cosmetic treatments; patients not likely to stay in the study for its duration because of other commitments, concomitant conditions, or past history; patients anticipated to be unreliable, or patients who have a concomitant condition that may develop symptoms that might confuse or confound study treatments or assessments).
   * Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alqam M, Wamsley CE, Hitchcock TM, Jones BC, Akgul Y, Kenkel JM. Efficacy and tolerability of a microneedling device for treating wrinkles on the face. J Cosmet Dermatol. 2023 Jan;22(1):206-213. doi: 10.1111/jocd.14985. Epub 2022 Jun 2. PMID 35403786

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre-screening was conducted by phone to determine eligibility criteria through an IRB-approved script. Followed by in-clinic screening visits conducted between
Pre-assignment Details: Only participants who met eligibility requirements were enrolled into the study.
  The subjects were given Pre-study instructions that include wash out Period: No topical medications or topical retinoids 2 weeks prior to visit 1.
Groups:
- Skinpen Precision System: Microneedle treatment to neck areas using SkinPen Precision system which includes: Surgical instrument motors and accessories/attachments/Hydrogel
  A total of 32 subjects completed study participation.
  At visit 1 (baseline), subjects were screened for eligibility criteria and those who qualified either completed day 1 procedures at the same visit or returned to the clinic up to 14 days after visit 1 to complete day 1 procedures at visit 2.
  On days 1, 30, 60, and 90, after completion of visit assessments, doctors or fellows at the testing facility (henceforth referred to as "clinic") treated each subject's fine lines and wrinkles, on the neck with SkinPen Precision System at depths of up to 2.5mm. Each subject's treatment depth was recorded. The hydrogel was used in conjunction with the treatment to protect against abrasion and friction during the procedure.
  During the treatment period (days 1-90), subjects used the supporting materials[SKINFUSE® Purify Cleansing Complex, Reclaim Hydrating Support (Moisturizer), and Shield Zinc Oxide Sunscreen] as directed.
Period: Overall Study
Arm/Group | Skinpen Precision System
Started | 35
Completed | 32
Not Completed | 3
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: At visit 1 (baseline), subjects were screened for eligibility criteria and those who qualified either completed day 1 procedures at the same visit or returned to the clinic up to 14 days after visit 1 to complete day 1 procedures at visit 2.
  35 Subjects were analyzed using the Fitzpatrick wrinkle scale and their scores are recorded.
Groups:
- SkinPen Precision System: Microneedle treatment to neck areas using SkinPen Precision system: Surgical instrument motors and accessories/attachments/Hydrogel.
  At visit 1 (baseline), subjects were screened for eligibility criteria and those who qualified either completed day 1 procedures at the same visit or returned to the clinic up to 14 days after visit 1 to complete day 1 procedures at visit 2.
  On days 1, 30, 60, and 90, after completion of visit assessments, doctors or fellows at the testing facility (henceforth referred to as "clinic") treated each subject's fine lines and wrinkles, on the neck with SkinPen Precision System at depths of up to 2.5mm. Each subject's treatment depth was recorded. The hydrogel was used in conjunction with the treatment to protect against abrasion and friction during the procedure.
  During the treatment period (days 1-90), subjects used the supporting materials[SKINFUSE® Purify Cleansing Complex, Reclaim Hydrating Support (Moisturizer), and Shield Zinc Oxide Sunscreen] as directed.
Arm/Group | SkinPen Precision System
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants] — Individuals deemed to have fine lines and wrinkles by the Investigator and that desire correction of their fine lines and wrinkles
  Participants
    <=18 years | 0
    Between 18 and 65 years | 35
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 3
Fitzpatrick Skin Classification [Number; unit: participants] — The Fitzpatrick skin classification is based on the skin's unprotected response to the first 30 to 45 minutes of sun exposure after a winter season without sun exposure. The categories of skin types are as follows:
  I-White, Always burns easily; never tans II-White, Always burns easily; tans minimally III-Cream white; Burns moderately; tans gradually IV-Brown; Mediterranean white skin. Burns minimally; always tans well V-Dark Brown; mid-eastern skin types, Rarely burns; tans profusely VI-Black; Never burns; deeply pigmented
  participants
    l | 0
    ll | 25
    lll | 5
    lV | 5
    V | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Wrinkle Severity Using the Lemperle Wrinkle Assessment Scale
Description: Wrinkling in the neck region will be assessed according to the following definitions:
  Class 0: No Wrinkles Class 1: Just perceptible wrinkle Class 2: Shallow wrinkles Class 3: Moderately deep wrinkle Class 4: Deep wrinkle, well-defined edges Class 5: Very deep wrinkle, redundant fold
Time Frame: Day 1 and 3 Month Post Treatment
Population: Analysis population includes all participants completing the study.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Skinpen Precision System: The subject's Fine lines and wrinkles were treated with the skinpen precision system at depths of 2.5mm. The hydrogel was used in conjunction with the treatment to protect against abrasion and friction during the procedure.
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 32
Score on a Scale
  Day 1 | 3.31 (0.74)
  3 Month Post Treatment | 2.45 (0.93)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using Wilcoxon signed rank test. Testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Clinician's Global Aesthetic Improvement Assessment (CGAIS)
Description: This scale is completed in two steps:
  * Based on a live assessment of the subject while referring to the subject's pre-treatment photographs of the neck, and
  * Based on a comparison of the subject's pre-treatment photographs to the current post-treatment photographs of the neck.
  Rating and its Description
  1 --Very Much Improved: Optimal cosmetic result in this subject. 2--Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal for this subject.
  3-Improved: Obvious improvement in appearance from the initial condition, but re-treatment is indicated.
  4--No Change: The appearance is essentially the same as the original condition. 5--Worse: The appearance is worse than the original condition.
Time Frame: 3 Month Post Treatment
Population: The analysis population includes all participants completing the study.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 32
Score on a Scale | 3.06 (0.74)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using Wilcoxon signed rank test. Testing hypothesis is that the mean score is equal to 4 (no change); Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Subject Global Aesthetic Improvement Scale (SGAIS)
Description: Rating and Description
  1. -Very Much Improved: Optimal cosmetic result.
  2. -Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal.
  3. -Improved: Obvious improvement in appearance from the initial condition.
  4. -No Change: The appearance is essentially the same as the original condition.
  5. -Worse: The appearance is worse than the original condition
Time Frame: 1 Month Post Treatment and 3 Month Post Treatment
Population: Analysis Population includes all participants completing the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 32
score on a scale
  1 Month Post Treatment | 2.90 (0.84)
  3 Month Post Treatment | 3.16 (0.72)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using the Wilcoxon signed rank test. Testing hypothesis is that the mean score is equal to 4; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Transepidermal Water Loss of the Left Neck by Biox Aquaflux
Description: The severity of wrinkles is more due to increased UV exposure through the driver's side window on the left side of the face and neck, due to this reason, the Principal investigator performed the TEWL on the left side of the neck. This test was pre-specified in the protocol. This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle.
  Biox Aquaflux is used to measure transepidermal water loss (TEWL) measurements which evaluate barrier function of the skin epidermal layer to determine the progress of epidermal healing after treatment.
  Day 1 will be used as a baseline to analyze the change from baseline. TEWL is measured in g/m2/h. Normal rates of TEWL - from 2.3 g/m2/h to 44 g/m2/h - are compromised due to injury, infection, and/or severe damage as in the case of burns A decrease inTEWL reflects less water loss and an improvement in the skin's barrier properties; an absence of a change in treate
Time Frame: Baseline, 3 Months post treatment
Population: Analysis population description includes all participants completing this test.
Measure: Mean (Standard Deviation); unit: g/m2/h
Arm/Group | SkinPen Precision System
Number analyzed (Participants) | 31
g/m2/h
  Baseline | 15.56 (6.72)
  3 Month post treatment | 14.62 (11.00)
Statistical Analysis 1: Comparison: SkinPen Precision System; Calculated using paired t-test. The testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p = 0.051, t-test, 1 sided

5. Secondary Outcome: Vascular Density Measurements by Optical Coherence Tomography(OCT)
Description: Vivosight, an Optical coherence tomography (OCT) device, is used to non-invasively gather topographical and histologic images of pre-and post-treated skin. This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle. OCT measurements of the vascular density are reported in percentage (%) and were performed on the neck at 100 microns, 200 microns, and 500 microns. Scores multiplied by 1000 for analysis.
  An increase in value indicates an increase in thickness and vascular density and skin tissue density.
Time Frame: Baseline (Day 1) and 3-Month post Treatment
Population: Analysis population includes everyone completing measurements art Baseline and 3 months post-treatment.
Measure: Mean (Standard Deviation); unit: % VD (Vascular Density)
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 31
% VD (Vascular Density)
  OTC Measure at 100 microns- Day 1 | 27.66 (19.76)
  OTC measure at 100 microns- 3 Month post treatment | 62.56 (55.97)
  OTC measure at 200 Microns- Day 1 | 74.45 (39.36)
  OTC measure at 200 Microns- 3 month Post treatment | 96.06 (56.25)
  OTC measure at 500 Microns- Day 1 | 45.81 (39.13)
  OTC measure at 500 Microns- 3 month Post treatment | 36.07 (40.91)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated from paired t-test. The testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p < 0.01, t-test, 1 sided

6. Secondary Outcome: Skin Roughness Measurements by Optical Coherence Tomography(OCT)
Description: Vivosight, an optical coherence tomography (OCT) device, was used to noninvasively gather topographical and histologic images of pre-and post-treated skin. This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle. Roughness measurements were calculated from the histologic images using RA and RZ. Skin roughness is measured in micro-meters.
  Ra is the average roughness of a surface. Rz is the difference between the tallest "peak" and the deepest "valley" on the surface.
  A decrease in value indicates a decrease in skin roughness when Baseline and 3 months post-treatment are compared.
Time Frame: Baseline (Day 1) and 3 Months post treatment
Population: The analysis population includes participants finishing this assessment at day 1 and 3 months post-treatment.
Measure: Mean (Standard Error); unit: micro-meters
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 25
micro-meters
  RA-Day 1 | 0.03 (0.04)
  RA-3 month post treatment | 0.01 (0.02)
  RZ-Day 1 | 0.11 (0.03)
  RZ- 3 Month Post treatment | 0.12 (0.05)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated from paired t-test. The testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p = 0.331, t-test, 1 sided

7. Secondary Outcome: BTC 2000 Measurements- Energy Absorption
Description: BTC-2000™ Features: High-Resolution Target Laser (µm) and negative pressure (mmHg & mbar)
  This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle.
  BTC 2000 was used to measure energy absorption of the skin.
  The units for these measurements are Energy absorption - mmHg*mm
  Decrease in values for energy absorption will be seen as Improvement
Time Frame: Baseline (Day 1) and 3 month post treatment
Population: Analysis population includes all participants completing this assessment on day 1 and 3 month post treatment.
Measure: Mean (Standard Deviation); unit: mmHg*mm
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 29
mmHg*mm
  Energy absorption-Day 1 | 105.78 (59.96)
  Energy absorption- 3 Month post treatment | 104.68 (65.86)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using the paired t test. Testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p = 0.863, t-test, 2 sided

8. Secondary Outcome: BTC 2000 Measurements for Skin Elasticity
Description: BTC-2000™ Features: High-Resolution Target Laser (µm) and negative pressure (mmHg & mbar)
  This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle.
  BTC 2000 was used to measure Elasticity values of the skin.
  The units for these measurements are in % of the distance traveled in µm.
  A decrease case in values for elasticity will be seen as an improvement after the treatments.
Time Frame: Baseline (Day 1) and 3 month post treatment
Population: Analysis population includes all participants completing this assessment on day 1 and 3 month post treatment.
Measure: Mean (Standard Deviation); unit: % of distance traveled in µm
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 29
% of distance traveled in µm
  Elasticity-Day 1 | 1.09 (0.60)
  Elasticity- 3 month post treatment | 5.33 (10.90)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using the paired t-test. The testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p = 0.048, t-test, 2 sided

9. Secondary Outcome: BTC 2000 Measurements for Skin Deformations
Description: BTC-2000™ Features: High-Resolution Target Laser (µm) and negative pressure (mmHg & mbar)
  This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle.
  BTC 2000 was used to measure viscoelastic deformation, elastic deformation, and ultimate deformation values of the skin.
  The units for these measurements are in mm.
  A Decrease in values for these deformations will be seen as an Improvement.
Time Frame: Baseline (Day 1) and 3 month post treatment
Population: Analysis population includes all participants completing this assessment on day 1 and 3 month post treatment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 29
mm
  Viscoelastic Deformation- Day 1 | 0.15 (0.11)
  Viscoelastic Deformation- 3 Month Post Treatment | 0.16 (0.13)
  Elastic Deformation- Day 1 | 2.44 (0.85)
  Elastic Deformation- 3 Month post treatment | 2.41 (0.87)
  Ultimate Deformation-Day 1 | 2.59 (0.95)
  Ultimate Deformation- 3 Month post treatment | 2.57 (0.96)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using the paired t-test. The testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p = 0.355, t-test, 2 sided — P-value reported is for viscoelastic deformation; at significance level alpha+0.05

10. Secondary Outcome: BTC 2000 Measurements for Stiffness
Description: BTC-2000™ Features: High-Resolution Target Laser (µm) and negative pressure (mmHg & mbar)
  This procedure was performed 4-6 cm from the left lateral neck along the sternocleidomastoid muscle.
  BTC 2000 was used for stiffness. Stiffness is measure in mmHg/mm and an increase in values of BTC measurements for stiffness would be seen as an improvement upon treatment.
Time Frame: Baseline (Day 1) and 3 month post treatment
Population: Analysis population includes all participants completing this assessment on day 1 and 3 month post treatment.
Measure: Mean (Standard Deviation); unit: mmHg/mm
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 29
mmHg/mm
  Stiffness- Day 1 | 165.24 (65.92)
  Stiffness- 3 Month Post treatment | 172.21 (65.18)
Statistical Analysis 1: Comparison: Skinpen Precision System; Calculated using the paired t test. Testing hypothesis is that the mean change from baseline is zero; Test type: Superiority; p = 0.859, t-test, 2 sided — Calculated with a paired T test. Testing hypothesis is that the mean change from baseline is zero

11. Secondary Outcome: Patient Satisfaction Questionnaires
Description: Subjects completed a Sponsor-provided questionnaire regarding improvement in wrinkles, satisfaction with the treatment, and willingness to recommend the treatment to friends and family members
Time Frame: 1 month post treatment
Population: All
Measure: Count of Participants; unit: Participants
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 32
Participants
  Do you notice any improvement in how your wrinkles look in the treated area?: Yes- 1 Month post treatment | 30
  Do you notice any improvement in how your wrinkles look in the treated area?: No-1 Month post Treatment | 2
  Reduction in the number of wrinkles: Yes- 1 Month post treatment | 12
  Reduction in the number of wrinkles: No-1 Month post Treatment | 20
  Reduction in the size of wrinkles: Yes- 1 Month post treatment | 25
  Reduction in the size of wrinkles: No-1 Month post Treatment | 7
  Reduction in Pore Size: Yes- 1 Month post treatment | 11
  Reduction in Pore Size: No-1 Month post Treatment | 21
  Clearer skin: Yes- 1 Month post treatment | 12
  Clearer skin: No-1 Month post Treatment | 20
  Smoother skin texture: Yes- 1 Month post treatment | 20
  Smoother skin texture: No-1 Month post Treatment | 12
  More even skin tone (color): Yes- 1 Month post treatment | 13
  More even skin tone (color): No-1 Month post Treatment | 19
  Would you recommend this treatment to your friends and family: number analyzed (Participants) | 31
  Would you recommend this treatment to your friends and family: Yes- 1 Month post treatment | 25
  Would you recommend this treatment to your friends and family: No-1 Month post Treatment | 6
Statistical Analysis 1: Comparison: Skinpen Precision System; Patient satisfaction questionnaires were tabulated, and the frequency and percentage of all response options were reported for each question and time point calculated from the binomial (sign) test. The testing hypothesis is that the proportion of favorable responses is equal to the unfavorable; Test type: Equivalence — .A binomial (sign) test was performed to test if the the proportion of the combined designated favorable evaluations/responses is equal to the combined designated negative evaluations/responses for each question; p < 0.01, Sign test

12. Secondary Outcome: Ultrasound Measurements
Description: Ultrasound measurements were performed using a 75 MHz ultrasonic transducer interfaced to a DUB 6100 OEM System (Taberna Pro Medicum, Lüneburg, Germany). Density and skin thickness measurements were obtained from the scans and increases in these values suggest a thickening of the epidermal and dermal tissue.
Time Frame: Day 1, 3 Months post treatment.
Population: The analysis population includes all participants completing this assessment.
Measure: Mean (Standard Deviation); unit: micro meter
Arm/Group | Skinpen Precision System
Number analyzed (Participants) | 26
micro meter
  Epidermal thickeness-Day 1 | 96.97 (52.99)
  Epidermal thickness-3 Month Post Treatment | 88.46 (26.21)
  Epidermal Density-Day 1 | 62.74 (23.28)
  Epidermal Density-3 M onth post treatment | 53.46 (24.22)
  Dermis Thickness-Day 1 | 1034.83 (247.72)
  Dermis Thickness- 3 Month Post treatment | 1092.08 (189.34)
  Dermis Density- Day 1 | 28.87 (13.67)
  Dermis Density- 3 Month Post treatment | 27.99 (15.01)
Statistical Analysis 1: Comparison: Skinpen Precision System; The null hypothesis that the mean change from baseline is zero was tested using a paired t-test; Test type: Superiority; p = 0.031, t-test, 2 sided — All statistical tests were 2-sided at significance level alpha=0.05. No multiple testing corrections were considered in the study

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from Baseline up to 6 months post treatment.
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation where a subject is administered any product or medical device, regardless of a causal relationship with the test article
Groups:
- Skinpen Precision System: Microneedle treatment to neck areas.
  SkinPen Precision: Surgical instrument motors and accessories/attachments/Hydrogel
Arm/Group | Skinpen Precision System
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 10/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skinpen Precision System (N=35)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Subject was in Follow up (not receiving treatment) when the AE was reported to the testing facility.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Kidney Stone removal (Renal and urinary disorders) | 1 (1)
Root canal (Gastrointestinal disorders) | 1 (1)
Meniscus repair (Gastrointestinal disorders) | 1 (1)
Sleep Apnea (Nervous system disorders) | 1 (1)
Biopsy on Jawline (Surgical and medical procedures) | 1 (1)
Viral Bronchitis (Infections and infestations) | 1 (1) — Subject was in Follow up (not receiving treatment) when the AE was reported to the testing facility.
Afib Cardioversion (Surgical and medical procedures) | 1 (1) — Subject was in Follow up (not receiving treatment) when the AE was reported to the testing facility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT03803059/Prot_SAP_000.pdf